CLINICAL TRIAL: NCT07322159
Title: An Exploratory Study of Safety and Efficacy of IASO206 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: IASO206 in Patients With Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025097
Record Dates: First submitted 2025-12-09; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IASO206 (Active Comparator): IASO206 will be administered in one infusion.
  Interventions: Drug: IASO206 injection

INTERVENTIONS:
Drug: IASO206 injection — The third-generation self-inactivating lentiviral vector that carries a BCMA-targeted CAR.

SUMMARY:
This study is an open-label, single-arm early exploratory clinical study, aiming to evaluate the safety, tolerability and preliminary efficacy of IASO206 Injection(In Vivo CAR-T) in Patients with Relapsed/Refractory Multiple Myeloma

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old, male or female;
* Diagnosed with relapsed/refractory multiple myeloma (RRMM) according to IMWG criteria, and have received at least 2 lines of treatment including one proteasome inhibitor and one immunomodulator; with documented disease progression (based on examination data) during or within 12 months after the latest anti-myeloma treatment (subjects whose last-line treatment was CAR-T therapy are not required to have progression within 12 months);
* Presence of measurable lesions during screening according to any of the following criteria:

  * Serum monoclonal protein (M-protein) level: ≥5 g/L f；
  * Urine M protein level ≥200 mg/24 hours;
  * Light chain multiple myeloma without measurable lesions in serum or urine: the affected serum free light chain ≥100 mg/L with abnormal serum κ/λ free light chain ratio;
* BCMA expression on MM cells determined by flow cytometry or pathology immunohistochemistry;
* ECOG score ≤ 2;
* Expected survival time ≥12 weeks;
* Subjects must have adequate organ function:
* Hematology: Absolute neutrophil count (ANC) ≥ 1×10^9/L (supportive treatment within 7 days before laboratory test is not allowed); Absolute lymphocyte count (ALC) )≥0.3×10^9/L; platelets≥50×10^9/L (blood transfusion support within 7 days before laboratory test is not allowed); hemoglobin ≥60 g/L (without red blood cell [RBC] transfusion within 7 days before laboratory test);

  * Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤1.5×upper limit of normal (ULN); serum total bilirubin≤1.5×ULN;
  * Renal function: creatinine clearance calculated according to Cockcroft-Gault formula≥ 40 ml/min.
  * Coagulation function: fibrinogen ≥1.0 g/L; activated partial thromboplastin time≤1.5×ULN, prothrombin time (PT)≤1.5×ULN;
  * Blood oxygen saturation>91%;
  * Left ventricular ejection fraction (LVEF) ≥50%;
* Subjects and their spouses agree to use effective contraceptive methods with tools or drugs from the time the subject signs the informed consent form until one year after administration;
* Subjects must sign a written informed consent form approved by the ethics committee before initiating the screening process.

Exclusion Criteria:

* Patients with suspected or confirmed central nervous system involvement by plasma cell neoplasms;
* Multiple myeloma patients with plasma cell leukemia;
* Patients with amyloidosis;
* Patients who have received autologous hematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks before enrollment, or have a history of allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
* Patients who have received previous BCMA-targeted therapy;
* Patients who have received plasma cell-targeted cellular therapy within 3 months before the screening period, or in whom received cellular therapy products can still be detected in peripheral blood;
* Patients who have received other anti-tumor treatments requires an appropriate washout period：

  * Received Bendamustine, fludalabine or high-dose cyclophosphoyl within 9 months before enrollment，or；
  * Received Monoclonal antibody treatment for multiple myeloma within 21 days before enrollment, or;
  * Received cytotoxic chemotherapy or proteasome inhibitor treatment within 14 days before enrollment, or；
  * Received immunomodulatory treatment within 7 days before enrollment, or;
  * Received other anti-tumor treatments (including but not limited to experimental drugs) listed above within 14 days before enrollment or at least 5 half-lives (whichever is longer);
* Patients requiring long-term use of therapeutic doses of corticosteroids during the study period (defined as prednisone or equivalent >20 mg/day), except for physiological replacement, topical, and inhaled use;
* Severe heart diseases：including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III), severe arrhythmia，hypertension that cannot be controlled by medication;
* Unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases；
* Patient who needs chronic use of immunosuppressive agents;
* Patients with malignant tumors other than multiple myeloma within 5 years before screening, excluding fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and those after radical resection Ductal carcinoma in situ of breast and papillary thyroid carcinoma;
* Patients with a history of solid organ transplantation;
* Major surgery history within 2 weeks before entering the study, or scheduled surgery during the study period or within 2 weeks after the study treatment；
* Serious uncontrolled infections during screening: Bacterial, viral, fungal, etc. infections;
* Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and detectable hepatitis B virus (HBV) DNA in peripheral blood; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus ( HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA test positive; syphilis test positive;
* Patients who have received inactivated vaccines within 4 weeks before enrollment;
* Women who are pregnant or breastfeeding;
* Patients with mental illness, consciousness disorder, or central nervous system diseases, including but not limited to epilepsy or a history of Parkinson's disease;
* Known severe allergic reaction to IASO206 or its formulation components (such as tocilizumab);
* Patients with unresolved non-hematological toxic reactions from previous treatments, which have not returned to baseline or ≤Grade 1 (except for alopecia and Grade 2 peripheral neuropathy);
* Other situations considered unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events（AEs） | up to 2 years after IASO206 infusion
  Cytokine release syndrome (CRS) and ICANS would be graded according to the ASTCT consensus.
  All other AEs would be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 2 years after IASO206 infusion
  The proportions of subjects achieving stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), and Partial Response (PR) after IASO206 infusion.
Time to response (TTR) | up to 2 years after IASO206 infusion
  The time from the start of the drug infusion in subjects to the first occurrence of sCR, CR, VGPR, or PR.
MRD negativity rate | up to 2 years after IASO206 infusion
  The proportion of subjects who achieve MRD-negativity after IASO206 infusion.
Duration of response (DOR) | up to 2 years after IASO206 infusion
  The time from the first assessment of sCR or CR or VGPR or PR to the first assessment of disease progression or death from any cause.
Progression-free survival (PFS) | up to 2 years after IASO206 infusion
  The time from the date IASO206 infusion to the date of first disease progression or death from any cause (whichever occurs first)
Overall survival (OS) | up to 2 years after IASO206 infusion
  The time from the date of IASO206 infusion to the date of death from any reason.
Pharmacodynamics（PD） | up to 2 years after IASO206 infusion
  The levels of cytokines (IL-6, serum ferritin, CRP) in peripheral blood at each time point，and lymphocyte subsets after IASO206 infusion.
Pharmacokinetic Analysis（PK） | up to 24 month after IASO206 infusion
  Maximum concentration (Cmax) of IASO206 particle and CAR-T cells.
Pharmacokinetic Analysis（PK） | up to 24 month after IASO206 infusion
  Time of maximum concentration (Tmax) of IASO206 particle and CAR-T cells.
Pharmacokinetic Analysis（PK） | up to 24 month after IASO206 infusion
  Area under the concentration versus time curve: IASO206 particle AUC0-12d; CAR-T cell AUC0-28d,AUC0-90d,AUC0-180d,AUC0-last

IPD SHARING:
Plan to Share IPD: No